CLINICAL TRIAL: NCT06373796
Title: Comparison of the Ultrasound Index Fat Fraction (FAT PLUS) With the MRI-PDFF Score for Quantification of Hepatic Steatosis.
Brief Title: Ultrasound Index Fat Fraction
Acronym: FAT-PLUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SuperSonic Imagine (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00523-44
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Steatosis of Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAT PLUS (Experimental)
  Interventions: Device: Echographic scan

INTERVENTIONS:
Device: Echographic scan — Liver ultrasound exam

SUMMARY:
The objective is to compare the ultrasound index fat fraction (FAT PLUS), derived from several ultrasound biomarkers, with the gold-standard imaging exam for liver fat content evaluation (MRI-PDFF) in patients to quantify the hepatic steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years old.
* Subject is able to understand and sign the Informed Consent Form.
* Subject is able to stand and walk independently.
* Subject must have at least one or more routine ultrasound imaging procedures of the abdomen, at one of the participating study sites.
* Subject must have at least one routine liver MRI with PDFF score performed within 30 days before or after the ultrasound examination
* Subject is affiliated to National Social Insurance or a Health Insurance Regimen

Exclusion Criteria:

* Subject is unable or unwilling to adhere to Study procedures
* Subject is unable to understand the Informed Consent
* Subject is unable to express its consent
* Subject is under legal protection
* Subject is deprived of liberty by judicial or administrative decision
* Subject undergoes psychiatric treatment under constraint
* Subject is pregnant or breastfeeding
* Subject has latex allergy
* Subject has an open wound, cut, and/or a rash which would preclude an ultrasound imaging procedure

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
FAT PLUS | 3 months
  The objective is to compare the ultrasound index fat fraction (FAT PLUS), derived from several ultrasound biomarkers, with the gold-standard imaging exam for liver fat content evaluation (MRI-PDFF) in patients to quantify the hepatic steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Aubé, MD, Principal Investigator — University Hospital, Angers
Locations (1):
- CHU Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided